CLINICAL TRIAL: NCT03109587
Title: Pilot Study of Probiotics in Pre-diabetic Adolescents
Acronym: ProDP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Christian L Roth, MD, Professor, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Probiotics/Diabetes Prevention
Record Dates: First submitted 2017-03-27; First posted 2017-04-12 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study product will be prepackaged and will be supplied and labeled only with the Protocol Number.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vivomixx (Visbiome) (Active Comparator): 2 packets of probiotics by mouth/day for 12 weeks
  Interventions: Dietary Supplement: Vivomixx
- Placebo (Placebo Comparator): identical in appearance, but without probiotics.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vivomixx — 900 billion of the following probiotic strains: L. acidophilus DSM24735; L. plantarum DSM24730; L. paracasei DSM24733; L. delbrueckii supsp. bulgaricus DSM24734, S. thermophilus DSM24731, B. longum DSM24736, B. breve DSM24732, and B. infantis DSM24737) maltose (polysaccharide used as food additive, produced from starch), and silicon dioxide (food additive)
  Arms: Vivomixx (Visbiome)
Dietary Supplement: Placebo — maltose (polysaccharide used as food additive, produced from starch), and silicon dioxide (food additive)
  Arms: Placebo

SUMMARY:
This study evaluates the feasibility and effect of probiotics on glycemic control in obese adolescents.

DETAILED DESCRIPTION:
Diet-induced intestinal dysbiosis in obese children contributes to the development of type 2 diabetes mellitus (T2D). Probiotic treatment has been proposed to alleviate glycemic dysfunction and prevent/delay development of T2D. The investigators will test probiotics to improve insulin sensitivity and preserve beta cell function in obese children.

The probiotic strains are known to improve glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 13-19 y. of age at Visit 1.
* BMI: 99th percentile or greater
* Acanthosis nigricans
* Pubertal Tanner stage ≥3

Exclusion Criteria:

* Secondary diabetes (i.e. post-transplant diabetes mellitus (DM) or cystic fibrosis DM), monogenic forms of diabetes (i.e. MODY), autoimmune diabetes or presence of islet autoantibodies.
* Known severe immunodeficiency, or immune compromised.
* Current or previous history for insulin or metformin therapy (within last 3 months).
* Antibiotic or probiotic therapy 3 months prior to enrollment.
* Start of new dietary intervention within 1 month prior to enrollment.
* Diagnosed food hypersensitivity or active gastrointestinal disease

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Change in microbiota composition | Baseline and 12 weeks
  Microbiome (16S rRNA) analysis, fecal immunoglobulin (Ig)A

SECONDARY OUTCOMES:
Change in insulin resistance | baseline and 12 weeks
  Measures of homeostatic model assessment of insulin resistance (HOMA-IR)
Change in inflammation in blood | baseline and 12 weeks
  measures of high sensitive cardio-reactive protein (hsCRP)
Change in inflammation in the gut | baseline and 12 weeks
  measure of fecal calprotectin

CONTACTS AND LOCATIONS:
Overall Officials: Christian L Roth, MD, Principal Investigator — Seattle Children's Hospital; Christiane S Hampe, PhD, Principal Investigator — University of Washington
Locations (1):
- Seattle Children's Hosptital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Verma A, Nelson MT, DePaolo WR, Hampe C, Roth CL. A randomized double-blind placebo controlled pilot study of probiotics in adolescents with severe obesity. J Diabetes Metab Disord. 2021 Aug 8;20(2):1289-1300. doi: 10.1007/s40200-021-00855-7. eCollection 2021 Dec. PMID 34900780